CLINICAL TRIAL: NCT05049603
Title: Phase III, Double-blinded, Multicenter, Randomized Clinical Trial to Evaluate the Effects of Atorvastatin on Moderate-to-severe and Active Graves' Orbitopathy (GO) Treated With Intravenous Glucocorticoids: the STAGO-2 Study
Brief Title: A Randomized Clinical Trial to Evaluate the Effects of Atorvastatin on Graves' Orbitopathy (GO): the STAGO-2 Study
Acronym: STAGO-2
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pisa (Other)
Collaborators: Università degli Studi dell'Insubria (Other); University of Catania (Other); University of Messina (Other)
Responsible Party: Principal Investigator, Marinò Michele, Associate Professor, University of Pisa
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STAGO-2
Record Dates: First submitted 2021-09-02; First posted 2021-09-20 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Graves' Orbitopathy
MeSH Terms: conditions — Graves Ophthalmopathy | interventions — Atorvastatin

STUDY DESIGN:
Intervention Model Description: Standard therapy (intravenous glucocorticoids) plus atorvastatin vs standard therapy plus placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study will be double-blinded. Investigational Pharmacy will prepare identical bottles containing the medications. Each bottle will be marked with a code, to be assigned to a patient. Once a patient is screened and eligible, upon request from Centers, Investigational Pharmacy will send sets of 2 bottles per patient (one containing atorvastatin and one containing placebo). Following randomization, the Investigational Pharmacy will communicate to the Center the code of the bottle to be used. On-site principal investigators will be entitled to identify a patient's intervention only in the case of an emergency. Data from patients collected in an online, password-protected, central database, will be handled by the statistician, who will perform the final analyses. The statistician will be informed the Investigational Pharmacy to which randomization group patients were assigned to, in order to perform the analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Atorvastatin (Experimental): Atorvastatin 20 mg/day (the experimental treatment), one tablet/day, given approximately at 10 pm, after dinner and before going to bed, for 24 weeks, associated with intravenous methylprednisolone pulse therapy (the standard treatment), given over a period of 12 weeks
  Interventions: Drug: Atorvastatin 20mg
- Placebo (Placebo Comparator): Intravenous methylprednisolone pulse therapy (the standard treatment), given over a period of 12 weeks, and placebo (one tablet/day, given approximately at 10 pm, after dinner and before going to bed) for 24 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Atorvastatin 20mg — One tablet/day, given approximately at 10 pm, after dinner and before going to bed, for 24 weeks
  Other Names: Study Group
  Arms: Atorvastatin
Other: Placebo — One tablet/day, given approximately at 10 pm, after dinner and before going to bed, for 24 weeks
  Other Names: Placebo group
  Arms: Placebo

SUMMARY:
Graves' orbitopathy (GO) is the most common extra-thyroidal manifestation of Graves' disease (GD). Based on its clinical signs and symptoms, GO is graded as mild, moderate-to-severe, or severe, and active or inactive, the latter feature being established on a 5/7-scale score named Clinical Activity Score (CAS).

The European Group on Graves Orbitopathy (EUGOGO) has recently formulated and published up-to-date guidelines for the management of GO, according to which high dose intravenous (iv) glucocorticoids (GC) (ivGC) is the first line treatment for moderate-to-severe and active GO. A protective effect of atorvastatin on the development of GO in patients with GD has been reported, based on which we recently conducted a phase II, randomized, open label clinical trial and found that atorvastatin improves the response of GO to ivGCs in hypercholesterolemic patients. The effect was unrelated to cholesterol levels, suggesting that it may be the consequence of a direct action of atorvastatin. To investigate this issue further and to introduce atorvastatin in the clinical practice, we designed the present Phase III, double-blinded, multicenter, randomized, adaptive, superiority, no profit, clinical trial to evaluate the effects of atorvastatin on Graves' Orbitopathy (GO) in patients with moderate-to-severe and active GO subjected to intravenous glucocorticoid therapy, regardless of cholesterol levels.

DETAILED DESCRIPTION:
Graves' orbitopathy (GO) is the most common extra-thyroidal manifestation of Graves' disease (GD). GO profoundly impairs the quality of life of affected patients. The pathogenesis is autoimmune, reflecting cross-reactivity against antigens shared by thyroid epithelial cells and orbital fibroblasts. Once the autoimmune reaction is initiated, a series of molecular mechanisms involving T and B cells, antibodies, cytokines, and oxidative stress, lead to fibroblast proliferation and release of glycosaminoglycans, resulting in the clinical manifestations of the disease, namely exophthalmos (or proptosis), soft tissue inflammation, diplopia, and in the most severe cases sight reduction or loss, due to corneal damage or to compression of the optic nerves, the so called optic neuropathy. Based on its clinical signs and symptoms, GO is graded as mild, moderate-to-severe, or severe, and active or inactive, the latter feature being established on a 5/7-scale score named Clinical Activity Score (CAS).

The European Group on Graves Orbitopathy (EUGOGO), a scientific Society involving several European Centers, including some of the Centers participating in the present study, has formulated and published up-to-date guidelines for the management of GO, which is referred to across the present study protocol.

According to EUGOGO guidelines, high dose intravenous (iv) glucocorticoids (GC) (ivGC) is the first line treatment for moderate-to-severe and active GO. The use of systemic glucocorticoids takes advantage from their immunosuppressive and anti-inflammatory actions, resulting in an overall beneficial effect ranging from ~35 to ~60% of patients in various studies. Recent studies have provided evidence for the best balance in terms of effectiveness/risks for a total methylprednisolone dose of 4.5 g, given in 12 weekly administrations, six of 500 and six of 250 mg, which is therefore recommended.

Besides genetic and demographical variables, risk factors associated with the development of GO in GD patients are known to be inadequate control of hyperthyroidism, radioiodine treatment, and smoking. In a large retrospective study conducted in more than 8,000 individuals with GD, it was reported that treatment with 3-hydroxy-3-methylglutaryl-coenzyme reductase inhibitors, better known as statins, especially atorvastatin, is associated with a ~40% reduced risk of developing GO in GD patients. The findings were interpreted as the consequence of the anti-inflammatory action of statins, being GO an autoimmune, inflammatory condition. Statins influence autophagic events and it has been shown that they induce cell death of human fibroblasts through a complex mechanism involving co-regulation of apoptosis, autophagy, and unfolded protein response (UPR). Thus, statins may reduce GO risk by modulating both apoptosis and autophagy activities. The molecular mechanisms that determine autophagy, apoptosis, and their interaction are not fully established, but the impact of statins on these two processes and their interplay in different cell types may provide a novel explanation for their pleiotropic effects in GO. Shih et al. found a positive correlation between macrophage count in the Muller's muscle and severity of upper lid retraction and concluded that the degree of inflammatory cell infiltration of Muller's muscle is associated with clinical severity of upper eyelid retraction in GO. Because some statins potently affect macrophage viability in vitro through the induction of apoptotic process, it is plausible that the early autophagic flux induced by statin treatment may be a potential mechanism to induce apoptosis of Muller's muscle infiltrating macrophages in patients with GO, thus eliciting a beneficial effect.

In addition to a possible direct action of statins on the eye, the possibility exists that the action of statins in GO may additionally reflect lowering of cholesterol. Thus, in a recent cross-sectional study a direct correlation between total and LDL-cholesterol levels and the presence and activity of GO in unselected patients with a GD of recent onset was observed, suggesting a direct link between cholesterol and GO. In addition, LDL-cholesterol was found to be a predictor of response to treatment. The mechanisms responsible for the relation between the presence of GO and cholesterol may be related to the altered inflammatory state of hypercholesterolemia. Thus, it is well known that disorders of lipid metabolism are associated with a state of mild-to-moderate, systemic, chronic inflammation. The increase load of free fatty acids on the liver, present in hyperlipemic states, causes dysfunction of the mitochondria and endoplasmic reticulum of hepatocytes, leading to the release of reactive oxygen radical species. In addition, free fatty acid can indirectly cause the release of pro-inflammatory cytokines, namely interleukin-6 and tumor necrosis factor-α, both involved in the pathogenetic mechanisms of GO.

Based on these findings, the investigators recently conducted a phase II, randomized, open label, external ophthalmological investigator-blinded, pilot, clinical trial, to determine whether administration of statins increases the efficacy of ivGC in patients with moderate-to-severe, active GO. Atorvastatin improved the response of GO to ivGCs in hypercholesterolemic patients. The effect was unrelated to cholesterol levels, suggesting that it may be the consequence of a direct action of atorvastatin. To investigate this issue further and to introduce atorvastatin in the clinical practice, the present Phase III, double-blinded, multicenter, randomized, adaptive, superiority, no profit, clinical trial was designed to evaluate the effects of atorvastatin on Graves' Orbitopathy (GO) in patients with moderate-to-severe and active GO subjected to intravenous glucocorticoid therapy, regardless of cholesterol levels.

ELIGIBILITY:
Inclusion Criteria

1. Patients willing and capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form
2. A diagnosis of Graves' disease based on the presence of hyperthyroidism associated with detectable anti-thyrotropic hormone (TSH) receptor autoantibodies (TRAb). Patients must be euthyroid under control on stable medical regimen and every effort will be made to maintain the euthyroid status for the entire duration of the clinical trial
3. A moderate-to-severe GO, defined as the presence of at least one of the following criteria: an exophthalmos ≥2 mm compared with normal values for sex and race; presence of inconstant to constant diplopia; a lid retraction ≥2 mm, lasting since no longer than 9 months
4. Active GO: CAS (4) ≥ 3 out of 5 points in the most affected eye
5. Male and female patients of age: 18-75 years
6. AST, ALT and CPK levels ≤ 3 times the upper value of normal range
7. Women of childbearing potential (WOCBP, namely not in menopause or in menopause since less than two years; in all other instances women will be considered as non-WOCBP) and men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year (as indicated in Appendix) for at least 6 and 7,5 months, respectively, after the last dose of the investigational drug (see also 2014_09_HMA_CTFG_Contraception.pdf, namely the "2014 CTFG Reccommendtions related to contraception and pregnancy testing in clinical trials").
8. Compliant patient, regular follow-up possible

Exclusion Criteria

1. Optic neuropathy
2. Corticosteroids or immunosuppressive treatment for GO in the last 3 months. Use of selenium in the last 3 months or during the clinical trial
3. Previous surgical or radiant (orbital irradiation) treatment for GO
4. Radioiodine treatment for hyperthyroidism over the last 3 months, as it can affect GO (4)
5. Statin treatment in the last 3 months
6. Contraindications to GC: hypersensitivity to the active substance or to any of the excipients; uncontrolled hypertension, uncontrolled diabetes; history of peptic ulcer; urinary infections, glaucoma, systemic fungal infections, systemic infections unless appropriate therapy is employed, idiopathic thrombocytopenic purpura, cerebral edema associated with malaria. Use of medications interfering with GC or increasing the risk of GC-related adverse events (see prohibited therapies)
7. Pregnant or lactating females as determined by positive serum or urine HCG test at baseline
8. Acute or chronic liver disease
9. All factors that could increase the risk of rhabdomyolysis, in particular medications that could increase this risk (see prohibited therapies)
10. Contraindications to statins, namely: hypersensitivity to atorvastatin or other statins, or hypersensitivity or intolerance to the medication excipients such as lactose; current or past liver diseases; alterations of liver tests.
11. Medications interfering/interacting with statins (see prohibited therapies)
12. Relevant Malignancy
13. Recent (≤1 year) history of alcoholism or drug abuse
14. Mental illness that prevent patients from comprehensive, written informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Outcome of GO | 24 weeks
  Comparison of overall GO outcome determined using a composite evaluation (% of responders).
  Response is defined as change in two outcome measures in at least one eye, without deterioration in any of the same measures in both eyes (compared to baseline):
  Patients meeting the improvement criteria will be considered as "responders". All other patients will be considered as "non-responders".

SECONDARY OUTCOMES:
Outcome of GO | 12 weeks
  Comparison of overall GO outcome determined using a composite evaluation (% of responders).
  Response is defined as change in two outcome measures in at least one eye, without deterioration in any of the same measures in both eyes (compared to baseline):
  Patients meeting the improvement criteria will be considered as "responders". All other patients will be considered as "non-responders".
Outcome of GO | 48 weeks
  Comparison of overall GO outcome determined using a composite evaluation (% of responders).
  Response is defined as change in two outcome measures in at least one eye, without deterioration in any of the same measures in both eyes (compared to baseline):
  Patients meeting the improvement criteria will be considered as "responders". All other patients will be considered as "non-responders".
Quality of life (comparison between the two groups) | 12 weeks
  Quality of life (QoL) will be evaluated using the GO QoL questionnaire (GO-QoL). Questionnaire consists of two subscales: 1) visual functioning (eight questions concerning limitations attributable to decreased visual acuity, diplopia, or both), and 2) appearance (eight questions referring to limitations in psychosocial functioning attributable to changes in appearance). Questions are scored as severely limited (one point), a little limited (two points), or not limited at all (three points). The two scores (8-24 points) are summed into a total score. A higher score means a better QoL. The total score and the subscores will be compared between the two groups
Quality of life (comparison between the two groups) | 24 weeks
  Quality of life (QoL) will be evaluated using the GO QoL questionnaire (GO-QoL). Questionnaire consists of two subscales: 1) visual functioning (eight questions concerning limitations attributable to decreased visual acuity, diplopia, or both), and 2) appearance (eight questions referring to limitations in psychosocial functioning attributable to changes in appearance). Questions are scored as severely limited (one point), a little limited (two points), or not limited at all (three points). The two scores (8-24 points) are summed into a total score. A higher score means a better QoL. The total score and the subscores will be compared between the two groups
Quality of life (comparison between the two groups) | 48 weeks
  Quality of life (QoL) will be evaluated using the GO QoL questionnaire (GO-QoL). Questionnaire consists of two subscales: 1) visual functioning (eight questions concerning limitations attributable to decreased visual acuity, diplopia, or both), and 2) appearance (eight questions referring to limitations in psychosocial functioning attributable to changes in appearance). Questions are scored as severely limited (one point), a little limited (two points), or not limited at all (three points). The two scores (8-24 points) are summed into a total score. A higher score means a better QoL. The total score and the subscores will be compared between the two groups
GO relapse | 24 weeks
  Worsening in comparison with the 12 week evaluation (% of relapse)
  Worsening is defined as change in two outcome measures in at least one eye (compared to 12 week):
GO relapse | 48 weeks
  Worsening in comparison with the 12 week evaluation (% of relapse)
  Worsening is defined as change in two outcome measures in at least one eye (compared to 12 week):

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Cisanello-Endocrinology II, Pisa, Italy

IPD SHARING:
Plan to Share IPD: No